CLINICAL TRIAL: NCT01590199
Title: Extension Study to the "Open-label Phase I Study Evaluating the Safety and Tolerability of Pasireotide LAR in Combination With Everolimus in Advanced Metastatic NETs - The COOPERATE-1 Study"
Brief Title: Evaluate Safety and Tolerability of Pasireotide LAR in Combination With Everolimus in Advanced Metastatic NETs
Acronym: MACS2002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001KDE47
Record Dates: First submitted 2012-04-11; First posted 2012-05-02 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Everolimus; pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RAD001 + SOM230 (Experimental)
  Interventions: Drug: RAD001; Drug: SOM230

INTERVENTIONS:
Drug: RAD001
  Other Names: Everolimus
Drug: SOM230
  Other Names: Paseriotide

SUMMARY:
This study will evaluate long-term safety and tolerability of pasireotide LAR in combination with everolimus in advanced metastatic NET patients, who who have not progressed during 12 months of combination therapy with pasireotide LAR and everolimus

ELIGIBILITY:
Inclusion and Exclusion Criteria:

Patients eligible for inclusion in this extension study have to meet all of the additional inclusion criteria:

* The patient must provide a signed Informed Consent Form (ICF) for the extension study prior to any study related procedures
* Completion of the whole treatment period of 15 months (3 months monotherapy with either pasireotide LAR or everolimus followed by a 12 months combination of pasireotide LAR/everolimus) in the CSOM230F2102 study
* No tumor progression during 12 months of combination therapy with pasireotide LAR and everolimus (checked via radiologically assessment).

No intolerable toxicity during combination therapy with pasireotide LAR and everolimus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-05-18 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events and Serious Adverse Enents as a Measure of Safety and Tolerability | up to 4 years
Number of Participants with abnormal laboratory and ECG results as a Measure of Safety and Tolerability | up to 4 years

SECONDARY OUTCOMES:
investigator-assessed progression free survival (PFS) | up to 4 years
best overall response | up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Germany (3):
  - Novartis Investigative Site, Bad Berka
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Münster

IPD SHARING:
Plan to Share IPD: Undecided